CLINICAL TRIAL: NCT05244590
Title: Development and Evaluation of a Mix-method Intervention Involving Training and a New Consultation Model for Patients With Palliative Care Needs in Primary Care - Before-After Study
Brief Title: Primary Care Consultation for Patients With Palliative Care Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Carlos Seiça Cardoso, Primary investigator, University of Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007015580
Record Dates: First submitted 2022-02-04; First posted 2022-02-17 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Palliative Care; Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): GPs' eligibility criteria
  * Working in the centre health care region in Portugal.
  * Authorisation of the coordinator of each GP health care unit to integrate the study.
  Patients' eligibility criteria
  Inclusion criteria
  * Belonging to the list of patients of the recruited GPs.
  * 18 years or older.
  * Diagnosis of advanced stage neoplasm (ASN), Chronic Obstructive Pulmonary Disease (COPD) Gold III/IV, Congestive Heart Failure (CHF) NYHA III/IV, Chronic Kidney Disease (CKD) stage IV/V.
  Exclusion Criteria
  * Refusal, at any time, to participate in the study.
  * Level of understanding or execution that compromises taking part in the study and answering the IPOS patient version (evaluated using Mini Mental State Examination score).
  * Level of disease severity requiring urgent intervention (GP clinical judgement).
  Interventions: Other: Consultation model for patients with palliative care needs

INTERVENTIONS:
Other: Consultation model for patients with palliative care needs — Training in PC for GPs The training program for GPs will meet the main training needs of GPs according to our previous study and feedback from elements of the Palliative Care Study Group of the Portuguese Association of General and Family Medicine (GESPal). The training program will have a total duration of 24 hours and will consist of two modules.
  Consultation model for patients Consultations will take place every 3 weeks for a total period of 12 weeks. The consultation model will be divided into five areas (Summarize clinical information, Objective symptoms' management, Assessment and coding of chronic diseases and symptoms, planning clinical approach, (other) problems/concerns) to be addressed during the assessment. The five areas were constructed to be intuitive for GPs, following the records' structure used in Portuguese primary care.

SUMMARY:
Introduction General practitioners provide health care in the community, managing patients and families longitudinally, and there is some evidence that when they are involved in caring for people with palliative care needs alongside specialists, palliative care delivery may be more efficient. The investigators aim to determine the impact of a mix-method intervention involving training in PC and a new consultation model for patients with palliative care needs in primary care.

Methods and analysis A before-after study will be conducted in the centre health care region of Portugal. The study will involve 53 patients with palliative care needs from the list of patients of the GPs who accept to collaborate with the project. The mix-method intervention will consist of: (1) training in palliative care and (2) application of a newly developed consultation model for use in the primary care setting and consisting of medical consultation every 3 weeks for a period of 12 weeks. The primary outcome is physical symptom burden, evaluated by the Integrated Palliative Outcome Scale (IPOS) patient version. Secondary outcomes include psychological symptoms, and communication/practical issues (IPOS); number of consultations for acute disease both in the health care unit and emergency department, number of hospitalizations and referrals to hospital health care services.

DETAILED DESCRIPTION:
Study aim:

The investigators aim to develop, apply, and evaluate a mix-method intervention involving training in PC and a new consultation model in primary care for patients with PC needs.

Primary objective:

To determine the impact of the intervention on the physical symptom burden for patients.

Secondary objectives:

To determine the impact of the intervention on:

1. psychological symptoms burden.
2. communication/practical issues.
3. some determinants of health care service use (number of consultations for acute disease both in the health care unit and emergency department, number of hospitalizations and referrals to hospital health care services).

Study design:

Before-after study

Study procedures:

GPs working in the centre health care region in Portugal will be asked to collaborate with the project.

GPs will receive a training program on PC built based on our previous study with GPs where the investigators identified the role of GPs in the PC setting and their training needs in PC. They will also receive training on how to apply the new consultation model.

Each GP will be asked to recruit patients with PC needs from their own list of patients using a protocol developed for that purpose. Each patient recruited will receive a medical consultation every 3 weeks for a period of 12 weeks. In both the first and last medical consultations, each GP will ask patients to complete the Integrated Palliative Outcome Scale (IPOS) patient version.

The study will integrate a pilot evaluation involving the first two patients of each GP, so that the consultation model can be improved according to the collected feedback.

The investigators intend to assess whether our mix-method intervention can improve the physical symptom burden of patients with PC needs after a 12-week intervention

Sample size:

Sample size was calculated for the main outcome (physical symptom burden) measured using the IPOS, considering the two time points (baseline and 12 weeks after). The effect of the intervention will be measured by the difference between the two means tested using t-test for paired samples, A sample size of 53 patients is estimated, considering a power of 80%, a type I error of 5%, and a medium effect size of 0.513, and accommodating a 50% loss of patients at follow-up (UCSF Clinical & Translational Science Institute - Sample Size Calculators, available at http://www.sample-size.net). Given that the prevalence of patients with PC needs in primary care is 8% to 14%3,4 and that in Portugal each GP has, on average, 1600 to 1900 patients in their list, it is estimated that each GP will have around 128 patients with PC needs in their list. Considering the involvement of 8-10 GPs in the study, the planned sample size is feasible. Included GPs will be asked to recruit patients until the planned sample size is reached (around 6 patients per GP).

Data collection:

The following variables will be collected by the main researcher about the GPs participating in the study: age, sex, years of clinical practice, type of primary care unit in which they work, environment (rural or urban) and previous training in PC.

The following variables will be collected by each GP about the patients participating in the study using a paper form: age, sex, education, marital status, rural or urban environment, main diagnosis, and comorbidities and IPOS patient version scores. GPs will also collect, by searching patients' medical records: number of consultations for acute disease both in the health care unit and emergency department, number of hospitalizations and referrals to hospital health care services referring to 12-week pre intervention and 12-week post intervention. A 12-week timeframe for evaluating resource use before and after the intervention was chosen to assess how these variables behaved over a period equal to that of the intervention. Each form will be pseudo-anonymized by assigning a code, so that only each GP will be able to identify which patient each form belongs to.

Statistical analysis:

Data analysis will be performed using SPSS v. 27®. Categorical variables will be described by frequencies (absolutes and relatives). Normally distributed continuous variables will be summarized by mean and standard deviation. Ordinal and non-normally distributed continuous variables will be represented by median and interquartile interval. The normality of the distributions will be assessed by observation of the respective QQ-plots.

To compare the difference of the two moments (baseline and 12 weeks after) a t-test for paired samples or a Wilcoxon test will be used. Statistical significance will be set at p<0.05.

ELIGIBILITY:
GPs' eligibility criteria Inclusion criteria

* Working in the centre health care region in Portugal.
* Authorisation of the coordinator of each GP health care unit to integrate the study.

Patients' eligibility criteria Inclusion criteria

* Belonging to the list of patients of the recruited GPs.
* 18 years or older.
* Diagnosis of advanced stage neoplasm (ASN), Chronic Obstructive Pulmonary Disease (COPD) Gold III/IV, Congestive Heart Failure (CHF) NYHA III/IV, Chronic Kidney Disease (CKD) stage IV/V.

Exclusion Criteria

* Refusal, at any time, to participate in the study.
* Level of understanding or execution that compromises taking part in the study and answering the IPOS patient version (evaluated using Mini Mental State Examination score).
* Level of disease severity requiring urgent intervention (GP clinical judgement).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Impact of the intervention in patients' physical symptom burden evaluated using Integrated Palliative Outcome Scale (IPOS) - patient version's mean scores | 12 week
  GPs enrolled will evaluate physical symptoms burden before and after the 12 week intervention.

SECONDARY OUTCOMES:
Impact of the intervention in patients' psychological symptoms burden evaluated using Integrated Palliative Outcome Scale (IPOS) - patient version's mean scores | 12 week
  GPs enrolled will evaluate psychological symptoms burden before and after the 12 week intervention.
Impact of the intervention in patients' communication/practical issues evaluated using Integrated Palliative Outcome Scale (IPOS) - patient version's mean scores | 12 week
  GPs enrolled will evaluate communication/practical issues before and after the 12 week intervention.
Impact of the intervention on number of consultations for acute disease both in the health care unit and emergency department, number of hospitalizations and referrals to hospital health care services | 12 week
  GPs enrolled will evaluate this variables 3 month before and 3 month after the 12 week intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- ARS Centro, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in peer-reviewed journals and presented at national and international conferences.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When the data is available

REFERENCES:
- [Derived] Seica Cardoso C, Prazeres F, Nunes C, Simoes P, Aires C, Rita P, Penetra J, Lopes P, Alcobia S, Gomes B. Impact of a complex intervention in primary care for patients with palliative care needs in their healthcare utilization: a before-after study. Prim Health Care Res Dev. 2026 Jan 30;27:e15. doi: 10.1017/S1463423625100777. PMID 41612825
- [Derived] Seica Cardoso C, Prazeres F, Oliveiros B, Nunes C, Simoes P, Aires C, Rita P, Penetra J, Lopes P, Alcobia S, Baptista S, Venancio C, Gomes B. Feasibility and effectiveness of a two-tiered intervention involving training and a new consultation model for patients with palliative care needs in primary care: A before-after study. Palliat Med. 2024 Sep;38(8):842-852. doi: 10.1177/02692163231219682. Epub 2024 Jan 16. PMID 38226491